CLINICAL TRIAL: NCT04495192
Title: Clinical, Neurophysiological and Genetical Predictors of Consciousness Recovery and Functional Outcomes After Severe Acquired Brain Injuries
Brief Title: Predictors of Better Outcomes After Severe Acquired Brain Injuries
Acronym: FP-GCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Bahia Hakiki, Neurologist, MD, Ph D, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: 16606_OSS
Record Dates: First submitted 2020-07-17; First posted 2020-07-31 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Brain Injuries; Disorder of Consciousness
Keywords: Rehabilitation; Machine Learning; Brain-derived neurotrophic factor; Apolipoprotein E; Cognitive Reserve; Predictive Factors
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders | interventions — Brain-Derived Neurotrophic Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by severe Acquired Brain Injury: All patients admitted in the participant IRU with a history of sABI and fulfilling our inclusion and exclusion criteria will be recruited.
  Interventions: Genetic: Genetic analysis of different single nucleotide polymorphisms on ApoE, BDNF and DRD2 genes assessment

INTERVENTIONS:
Genetic: Genetic analysis of different single nucleotide polymorphisms on ApoE, BDNF and DRD2 genes assessment — Genomic DNA will be obtained from EDTA-whole venous blood sample by Automated Systems QiaCube (Qiagen). The genetic analysis of 5 different single nucleotide polymorphisms on ApoE, BDNF and DRD2 genes will be performed by HRM analyses and direct sequencing on Automatic Genetic Analyzer. All the aliquots will be amplified by a real-time PCR. The genetic polymorphism data will be compared to sex- and age-matched control of the DNA banking of the neurogenetic Laboratory of Florence Hospital.

SUMMARY:
Severe Acquired Brain Injury is defined as a traumatic, post-anoxic, vascular or other brain damage that causes coma for at least 24 hours and leads to permanent disability with sensorial, motor, cognitive or compartmental impairment. In this context, an accurate characterization of individual patients' profile in terms of neuronal damage, potential for neuroplasticity, neurofunctional and clinical state could allow to plan tailored rehabilitation and care pathway on the basis of solid prognostic information, also for optimizing resources of the National Health care systems and enhance ethical decisions. Patient profiling should encompass measures and procedures easily available at the bedside, and with affordable time, resource, and money-costs to determine a real impact on National Health systems. The aim of the study is identifying patient profiles in terms of clinical, neurophysiological and genetical aspects with better long-term outcome in order to plan tailored therapeutic interventions.

DETAILED DESCRIPTION:
Background:

After a severe Acquired Brain Injury (sABI) the consciousness, the functional and the cognitive recovery of the patients depends on the severity of the damage suffered but also on the vulnerability of the individual brain. Some patients with sABI may survive in a state of Disorder of Consciousness (DoC) condition (i.e., patients in vegetative state/unresponsive wakefulness syndrome, VS/UWS or in minimally conscious state, MCS). Other patients, despite having a complete recovery of consciousness, can reach very variable degrees of functional and cognitive autonomy. The prognostic factors of consciousness recovery of patients with DoCs have been thoroughly investigated. Most of these studies investigated the acute phase, while only a few studies have examined the role of early clinical factors emerging before the complete recovery of consciousness . Further prognostic insights can be provided by analysis of genes coding for Apolipoprotein E (APOE), dopamineD2 receptor (DRD2), and Brain Derived Neutrophic Factors (BDNF), and by markers of axonal injury.

Study aim:

The present project aims at identifying patient profiles with better long-term outcome in order to plan tailored therapeutic interventions.

The patient profiles will be drawn up by gathering patient's demographic (age, gender, social and educational level), anamnestic (aetiology and time post-brain injury, Cognitive Reserve Index), clinical state (Cumulative Illness Rating Scale (CIRS), CRS-R total score and corresponding consciousness state; Disability Rating Scale, DRS, Functional Oral Intake Scale; FOIS, Glasgow Outcome Scale Expanded; GOS-E, Level of Cognitive Functioning; LCF) and neurophysiological data (Electroencephalogram (EEG), Somatosensory evoked potentials (SEP), and Motor evoked potentials (MEP) nerve conduction aimed at evaluating occurrence of critical illness polyneuropathy and myopathy (CIPNM)) at study entry (baseline), together with neural biomarkers (genetic markers).

On the basis of the above mentioned stratification of patients by this multimodal approach, the present study aimed to

1. Investigate the possible association of certain profiles with the consciousness recovery at the time of discharge from the Intensive Rehabilitation Unit (IRU), at 1 year and 2 years from the acute event
2. Investigate the possible association of certain profiles with the functional outcomes at the time of discharge from the Intensive Rehabilitation Unit (IRU), at 1 year and 2 years from the acute event.
3. Investigate the possible association of certain profiles with the long-term cognitive profile and the level of familiar and social participation at 1 year and 2 years from the acute event.

Setting , population and methods:

The proposed study is a longitudinal multi-location prospective observational cohort study.

Four centers of the Don Carlo Gnocchi Foundation will participate (Florence, La Spezia, Milan and Sant'Angelo dei Lombardi and the neurogenetics laboratory of the University of Florence, Department of Medical and Experimental Sciences, Neurology). The enrollment phase will last 3 years (June 2020-June 2023). 520 patients with severe brain injury will be included (200 for the Florence and La Spezia units and 60 for the Milan and Sant'Angelo dei Lombardi units).

All patients admitted in the participant IRU with a history of sABI within 4 months, aged 18+, presenting a signed informed consent signature for the participation to the study and for the genetic analysis will be consecutively enrolled.

A multidimodal evaluation including clinical examinations and neurophysiological assessments will be performed by skilled professionals. The study foresees four steps in the late acute phase and two in the long-term phase: 1) at the study entry time (T0), 2) at three months from T0 (T1) 3) at 6 months from T0 (T2) 4) at discharge (T3) 5) at 12 months from the acute event (T4) 6) at 24 months from the acute event.

Clinical assessment including :

1. Consciousness assessment using CRS-R
2. Care severity profile: including the comorbidity assessed thought the Cumulative Illness Rating Scale (CIRS), the presence of medical devices, sepsis occurrence during the IRU stay, neurosurgery interventions, bedsores, epileptic event and other complications
3. Functional evaluation using the following scales: ERBI, GOS-E, DRS, FIM, PAINED pain scale, TCT, Ashworth, FOIS
4. Neurocognitive profile evaluation using the Galveston Orientation and Amnesia Test (GOAT), the Level of Cognitive Functioning (LCF) and the International Classification of Functioning, Disability and Health (ICF), ABS, AES and Cognitive Reserve Index (CRI)

Multimodal neurophysiological evaluation including:

1. Standard EEG recording at rest. EEG background activity and reactivity will be classified according to recently proposed diagnostic criteria for DoC and to American Clinical Neurophysiology Society Critical Care EEG Terminology.
2. Motor and sensory nerve conduction studies. Sensory nerve action potentials, and compound muscle action potentials (CMAP) will be evaluated. Muscular activity at rest and when possible during reflex contraction will be assessed.
3. PEM: Transcranial magnetic stimulation (TMS) will be performed according to the standard criteria of the International Federation of Clinical Neurophysiology. MEP will be recorded from abductor digiti minimi and tibialis anterior muscles and size of MEP measured as MEP/CMAP amplitude ratio.
4. Bilateral upper limb SEP will be recorded according to the International Federation of Clinical Neurophysiology. The presence or absence of N20/P25 cortical components will be evaluated.

Genetic assessment Genomic DNA will be obtained from EDTA-whole venous blood sample by Automated Systems QiaCube (Qiagen). The genetic analysis of 5 different single nucleotide polymorphisms on ApoE, BDNF and DRD2 genes will be performed by high resolution melt (HRM) analyses and direct sequencing on Automatic Genetic Analyzer. APOE genotypes will be investigated by HRM with two sets of PCR primers designed to amplify the regions encompassing rs7412 [NC_000019.9: g.45412079C>T] and rs429358 (NC_000019.9: g.45411941T>C). The samples with known ApoE genotypes, which had been validated by DNA sequencing, will be used as standard references. The genetic polymorphism data will be compared to sex- and age-matched control of the DNA banking of the neurogenetic Laboratory of Careggi Hospital of Florence.

Statistic analysis:

All collected data will be analyzed using a machine learning algorithm, creating, for each patient, a risk profile for the possible consciousness recovery and functional autonomy.

On the basis of the results of this study, partecipant will build on a "decision support tool" for future sABI patients afferent to the Intensive Rehabilitative Unit, in order to plan personalized rehabilitative and therapeutic interventions, allowing therefore an optimization of resources (costs and resources) for National Health Service

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with a history of severe Acquired Brain Injury within 4 months,
* aged 18+,
* signed informed consent signature for the participation to the study
* signed informed consent signature for the participation to for the genetic analysis

Exclusion Criteria:

* patients admitted with a history of severe Acquired Brain Injury more then 4 months
* Absence of informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe Acquired Brain Injuries admitted in the Intensive Rehabilitative Unit (IRU) of the four participant don Gnocchi Foundation Centers (Florence, La Spezia, Milano and Sant'Angelo dei Lombardi) fulfilling the inclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Consciousness recovery | 24 months
  The Consciousness recovery will be measured throught the italian version of the CRS-R performed for at least 5 time during one week to avoid a misdiagnosis due to consciousness fluctuations.Consciousness recovery is defined as CRS_R >23 and Improvement Responsiveness will be registred for patients transitioning from UWS to MCS or E-MCS, and from MCS to E-MCS.
Tracheostomy weaning | 24 months
  Tracheostomy weaning will be reported as a dichotomic variable: decannulated yes/no
Total oral feeding recovery | 24 months
  The swallowing severity will be assessed throught the Oral feeding recovery measured by Functional Oral Intake Scale (FOIS) scoring from 1 (severe dysphagia) to 7(absence of dysphagia). The outcome of "oral feeding recovery" corrispond to Functional Oral Intake Scale>4
Functional autonomy | 24 months
  Functional autonomy measured by Glasgow Outcome Scale Expanded scoring between 1 (death) and 8 (complete functional recovery). A good autonomy is defined for Glasgow Outcome Scale Expanded >4
Time to decannulation | 24 months
  In decannulated patients, time between admission in the IRU and decannulation will be reported

SECONDARY OUTCOMES:
Cognitive profile | 24 months
  The cognitive profile will be assessed firstly investigating the "post-event amnesia" by the Galveston Orientation & Amnesia Test. The date of "post-event amnesia" resolution will be reported when the Galveston Orientation & Amnesia Test score >75 for two consecutive days
Degree of social and occupational reintegration | 24 months
  Degree of social and occupational reintegration assessed by the Community Integration Questionnaire (CIQ). Minimum score is 10 and maximum score is 50. A higher score indicates a higher comunity integration
Subjective and Objective Quality Of Life | 24 months
  The Quality of Life after Brain Injury (QoLibri) scale allows to measure both the quality of life perceived by both the patient and the caregiver. Quality of Life after Brain Injury (QoLibri) scores are reported on a 0-100 scale.
  0=worst possible quality of life and 100=best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bahia Hakiki, MD, Phd, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi, Florence
Locations (1):
- IRCCS-don Gnocchi Foundation, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernat JL. Chronic disorders of consciousness. Lancet. 2006 Apr 8;367(9517):1181-92. doi: 10.1016/S0140-6736(06)68508-5. PMID 16616561
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Hirschberg R, Giacino JT. The vegetative and minimally conscious states: diagnosis, prognosis and treatment. Neurol Clin. 2011 Nov;29(4):773-86. doi: 10.1016/j.ncl.2011.07.009. PMID 22032660
- [Background] Amantini A, Grippo A, Fossi S, Cesaretti C, Piccioli A, Peris A, Ragazzoni A, Pinto F. Prediction of 'awakening' and outcome in prolonged acute coma from severe traumatic brain injury: evidence for validity of short latency SEPs. Clin Neurophysiol. 2005 Jan;116(1):229-35. doi: 10.1016/j.clinph.2004.07.008. PMID 15589201
- [Background] Cavinato M, Freo U, Ori C, Zorzi M, Tonin P, Piccione F, Merico A. Post-acute P300 predicts recovery of consciousness from traumatic vegetative state. Brain Inj. 2009 Nov;23(12):973-80. doi: 10.3109/02699050903373493. PMID 19831494
- [Background] Portaccio E, Morrocchesi A, Romoli AM, Hakiki B, Taglioli MP, Lippi E, Di Renzone M, Grippo A, Macchi C; Intensive Rehabilitation Unit Study Group of the IRCCS Don Gnocchi Foundation, Italy. Improvement on the Coma Recovery Scale-Revised During the First Four Weeks of Hospital Stay Predicts Outcome at Discharge in Intensive Rehabilitation After Severe Brain Injury. Arch Phys Med Rehabil. 2018 May;99(5):914-919. doi: 10.1016/j.apmr.2018.01.015. Epub 2018 Feb 8. PMID 29428346
- [Background] Portaccio E, Morrocchesi A, Romoli AM, Hakiki B, Taglioli MP, Lippi E, Di Renzone M, Grippo A, Macchi C. Score on Coma Recovery Scale-Revised at admission predicts outcome at discharge in intensive rehabilitation after severe brain injury. Brain Inj. 2018;32(6):730-734. doi: 10.1080/02699052.2018.1440420. Epub 2018 Feb 26. PMID 29482376
- [Background] Scarpino M, Lolli F, Hakiki B, Atzori T, Lanzo G, Sterpu R, Portaccio E, Romoli AM, Morrocchesi A, Amantini A, Macchi C, Grippo A; Intensive Rehabilitation Unit Study Group of the IRCCS Don Gnocchi Foundation, Italy. Prognostic value of post-acute EEG in severe disorders of consciousness, using American Clinical Neurophysiology Society terminology. Neurophysiol Clin. 2019 Sep;49(4):317-327. doi: 10.1016/j.neucli.2019.07.001. Epub 2019 Jul 18. PMID 31327535
- [Background] Lammi MH, Smith VH, Tate RL, Taylor CM. The minimally conscious state and recovery potential: a follow-up study 2 to 5 years after traumatic brain injury. Arch Phys Med Rehabil. 2005 Apr;86(4):746-54. doi: 10.1016/j.apmr.2004.11.004. PMID 15827927
- [Background] Katz DI, Polyak M, Coughlan D, Nichols M, Roche A. Natural history of recovery from brain injury after prolonged disorders of consciousness: outcome of patients admitted to inpatient rehabilitation with 1-4 year follow-up. Prog Brain Res. 2009;177:73-88. doi: 10.1016/S0079-6123(09)17707-5. PMID 19818896
- [Background] Estraneo A, Moretta P, Loreto V, Lanzillo B, Santoro L, Trojano L. Late recovery after traumatic, anoxic, or hemorrhagic long-lasting vegetative state. Neurology. 2010 Jul 20;75(3):239-45. doi: 10.1212/WNL.0b013e3181e8e8cc. Epub 2010 Jun 16. PMID 20554941
- [Background] Lipsky RH, Lin M. Genetic predictors of outcome following traumatic brain injury. Handb Clin Neurol. 2015;127:23-41. doi: 10.1016/B978-0-444-52892-6.00003-9. PMID 25702208
- [Background] Kim BR, Kim HY, Chun YI, Yun YM, Kim H, Choi DH, Lee J. Association between genetic variation in the dopamine system and motor recovery after stroke. Restor Neurol Neurosci. 2016 Nov 22;34(6):925-934. doi: 10.3233/RNN-160667. PMID 27689550
- [Background] Sorbi S, Nacmias B, Piacentini S, Repice A, Latorraca S, Forleo P, Amaducci L. ApoE as a prognostic factor for post-traumatic coma. Nat Med. 1995 Sep;1(9):852. doi: 10.1038/nm0995-852. No abstract available. PMID 7585199
- [Background] Lanzillotta A, Pignataro G, Branca C, Cuomo O, Sarnico I, Benarese M, Annunziato L, Spano P, Pizzi M. Targeted acetylation of NF-kappaB/RelA and histones by epigenetic drugs reduces post-ischemic brain injury in mice with an extended therapeutic window. Neurobiol Dis. 2013 Jan;49:177-89. doi: 10.1016/j.nbd.2012.08.018. Epub 2012 Aug 30. PMID 22971966
- [Background] Thelin EP, Nelson DW, Vehvilainen J, Nystrom H, Kivisaari R, Siironen J, Svensson M, Skrifvars MB, Bellander BM, Raj R. Evaluation of novel computerized tomography scoring systems in human traumatic brain injury: An observational, multicenter study. PLoS Med. 2017 Aug 3;14(8):e1002368. doi: 10.1371/journal.pmed.1002368. eCollection 2017 Aug. PMID 28771476
- [Background] Mateen BA, Hill CS, Biddie SC, Menon DK. DNA Methylation: Basic Biology and Application to Traumatic Brain Injury. J Neurotrauma. 2017 Aug 15;34(16):2379-2388. doi: 10.1089/neu.2017.5007. Epub 2017 Jun 28. PMID 28482743
- [Background] Scarpino M, Lolli F, Hakiki B, Lanzo G, Sterpu R, Atzori T, Portaccio E, Draghi F, Amantini A, Grippo A; Intensive Rehabilitation Unit Study Group of the IRCCS Don Gnocchi Foundation, Italy. EEG and Coma Recovery Scale-Revised prediction of neurological outcome in Disorder of Consciousness patients. Acta Neurol Scand. 2020 Sep;142(3):221-228. doi: 10.1111/ane.13247. Epub 2020 Apr 14. PMID 32219851
- [Derived] Hakiki B, Liuzzi P, Romoli AM, Draghi F, Maccanti D, De Nisco A, Burali R, Toci T, Grippo A, Scarpino M, Mannini A, Magliacano A, Estraneo A, Comanducci A, Navarro J, Tramonti C, Carli V, Balbi P, Macchi C, Cecchi F. Predictors of Recovering Full Consciousness: Results From a Prospective Multisite Italian Study. Eur J Neurol. 2025 Apr;32(4):e70138. doi: 10.1111/ene.70138. PMID 40275709
- [Derived] Draghi F, Pancani S, De Nisco A, Romoli AM, Maccanti D, Burali R, Grippo A, Macchi C, Cecchi F, Hakiki B. Implications of the Consciousness State on Decannulation in Patients With a Prolonged Disorder of Consciousness. Arch Phys Med Rehabil. 2024 Sep;105(9):1691-1699. doi: 10.1016/j.apmr.2024.05.006. Epub 2024 May 10. PMID 38734048